CLINICAL TRIAL: NCT04631601
Title: A Master Protocol Evaluating the Safety and Efficacy of Therapies for Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Safety and Efficacy of Therapies for Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Amgen made a business decision to discontinue all AMG 160 clinical trials. This decision is not related to safety.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190505; 2020-001305-23 (EudraCT Number)
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Acapatamab; HALF-LIFE EXTENDED (HLE) BITE; mCRPC; Metastatic Castration-resistant Prostate Cancer; 68; Gallium (68Ga)-prostate-specific membrane; antigen (PSMA)-11 positron emission; tomography(PET)/computed tomography (CT); and; 18; F-fluorodeoxyglucose (FDG) PET/CT; based response evaluation; Bispecific T cell Engager; BITE
MeSH Terms: conditions — Bites and Stings | interventions — enzalutamide; Androgen Receptor Antagonists; abiraterone; Cytochrome P-450 Enzyme System; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Acapatamab and Enzalutamide: Dose Exploration (Experimental): The dose-exploration part of the study will estimate the MTD/recommended phase 2 dose (RP2D) of Acapatamab in combination with enzalutamide.
  Interventions: Drug: Acapatamab; Drug: Enzalutamide
- Acapatamab and Enzalutamide: Dose Expansion (Experimental): Following dose exploration, dose expansion will be conducted to confirm the safety and tolerability of the selected dose and to further evaluate the efficacy of Acapatamab in combination with enzalutamide.
  Interventions: Drug: Acapatamab; Drug: Enzalutamide
- Acapatamab and Abiraterone: Dose Exploration (Experimental): The dose exploration part of the study will estimate the MTD/recommended phase 2 dose (RP2D) of Acapatamab in combination with abiraterone.
  Interventions: Drug: Acapatamab; Drug: Abiraterone
- Acapatamab and Abiraterone: Dose Expansion (Experimental): Following dose exploration, dose expansion will be conducted to confirm the safety and tolerability of the selected dose and to further evaluate the efficacy of Acapatamab in combination with abiraterone.
  Interventions: Drug: Acapatamab; Drug: Abiraterone
- Acapatamab and AMG 404: Dose Exploration (Experimental): The dose-exploration part of the study will estimate the MTD/RP2D of Acapatamab in combination with AMG 404.
  Interventions: Drug: Acapatamab; Drug: AMG 404
- Acapatamab and AMG 404: Dose Expansion (Experimental): Following dose exploration, dose expansion will be conducted to confirm the safety and tolerability of the selected dose and to further evaluate the efficacy of Acapatamab in combination with AMG 404.
  Interventions: Drug: Acapatamab; Drug: AMG 404
- AMG 404 Monotherapy (Active Comparator): AMG 404 monotherapy is being conducted to evaluate the preliminary anti-tumor activity of PD-1 inhibition in the mCRPC population.
  Interventions: Drug: AMG 404
- Acapatamab and Enzalutamide: Dose Expansion Asia Cohort (Experimental): Following dose exploration, dose expansion will be conducted in the Asia cohort at the combination MTD/RP2D determined in dose exploration to confirm the safety, tolerability and PK of Acapatamab in combination with enzalutamide for subjects in Asia.
  Interventions: Drug: Acapatamab; Drug: Enzalutamide
- Acapatamab and Abiraterone: Dose Expansion Asia Cohort (Experimental): Following dose exploration, dose expansion will be conducted in the Asia cohort at the combination MTD/RP2D determined in dose exploration to confirm the safety, tolerability and PK of Acapatamab in combination with abiraterone for subjects in Asia.
  Interventions: Drug: Acapatamab; Drug: Abiraterone
- Acapatamab and AMG 404: Dose Expansion Asia Cohort (Experimental): Following dose exploration, dose expansion will be conducted in the Asia cohort at the combination MTD/RP2D determined in dose exploration to confirm the safety, tolerability and PK of Acapatamab in combination with AMG 404 for subjects in Asia.
  Interventions: Drug: Acapatamab; Drug: AMG 404
- Acapatamab Monotherapy (Experimental): Acapatamab monotherapy is being conducted to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and efficacy of Acapatamab in subjects with mCRPC.
  Interventions: Drug: Acapatamab

INTERVENTIONS:
Drug: Acapatamab — Acapatamab will be administered as an intravenous (IV) infusion.
  Other Names: PSMA targeted therapy
  Arms: Acapatamab Monotherapy; Acapatamab and AMG 404: Dose Expansion; Acapatamab and AMG 404: Dose Expansion Asia Cohort; Acapatamab and AMG 404: Dose Exploration; Acapatamab and Abiraterone: Dose Expansion; Acapatamab and Abiraterone: Dose Expansion Asia Cohort; Acapatamab and Abiraterone: Dose Exploration; Acapatamab and Enzalutamide: Dose Expansion; Acapatamab and Enzalutamide: Dose Expansion Asia Cohort; Acapatamab and Enzalutamide: Dose Exploration
Drug: Enzalutamide — Enzalutamide will be administered orally.
  Other Names: Androgen receptor inhibitor
  Arms: Acapatamab and Enzalutamide: Dose Expansion; Acapatamab and Enzalutamide: Dose Expansion Asia Cohort; Acapatamab and Enzalutamide: Dose Exploration
Drug: Abiraterone — Abiraterone will be administered orally.
  Other Names: Cytochrome P450 (CYP)17 inhibitor
  Arms: Acapatamab and Abiraterone: Dose Expansion; Acapatamab and Abiraterone: Dose Expansion Asia Cohort; Acapatamab and Abiraterone: Dose Exploration
Drug: AMG 404 — AMG 404 will be administered as an intravenous (IV) infusion.
  Other Names: PD-1 inhibitor
  Arms: AMG 404 Monotherapy; Acapatamab and AMG 404: Dose Expansion; Acapatamab and AMG 404: Dose Expansion Asia Cohort; Acapatamab and AMG 404: Dose Exploration

SUMMARY:
This is a master protocol designed to evaluate the safety and efficacy of investigational therapies in participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a master protocol designed to evaluate the safety, tolerability, and maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) and efficacy of Acapatamab, in combination with enzalutamide, abiraterone, or the PD1 inhibitor AMG 404, AMG 404 monotherapy, as well as Acapatamab monotherapy, in participants with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
All parts

Inclusion Criteria:

* ≥ 18 years of age (or legal adult age within country)
* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Subjects with mCRPC with histologically or cytologically confirmed adenocarcinoma of the prostate
* Subjects should have undergone bilateral orchiectomy or should be on continuous androgen deprivation therapy with a gonadotropin releasing hormone agonist or antagonist (testosterone ≤ 50 ng/dL (or 1.7 nmol/L))

Exclusion Criteria:

* Central nervous system (CNS) metastases or leptomeningeal disease
* History or presence of clinically relevant CNS pathology
* Confirmed history or current autoimmune disease or other diseases requiring permanent immunosuppressive therapy
* Myocardial infarction, uncontrolled hypertension, unstable angina, cardiac arrhythmia requiring medication, and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months
* Prior treatment with a taxane for mCRPC
* Major surgery and/or Radiation within 4 weeks
* History or evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection unless agreed upon with medical monitor and meeting the following criteria:

  * Negative test for SARS-CoV-2 RNA by real time polymerase chain reaction (RT-PCR) within 72 hours of first dose of Acapatamab (or AMG 404 in Part 3)
  * No acute symptoms of COVID-19 disease within 10 days prior to first dose of Acapatamab (or AMG 404 in Part 3) (counted from day of positive test for asymptomatic subjects)

Prior/Concurrent Clinical Study Experience

* Currently receiving treatment in another investigational device or drug study, or less than 4 weeks since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded with the exception of investigational scans.

Subprotocol A only:

Inclusion criteria

• Subjects planning to receive enzalutamide for the first time for mCRPC

Exclusion criteria

* Use of strong CYP2C8 inhibitors or strong CYP3A4 inducers
* Use of narrow therapeutic index drugs that are substrates of CYP3A4, CYP2C9 or CYP2C19

Subprotocol B only:

Inclusion criteria

* Subjects planning to receive abiraterone for the first time for mCRPC Exclusion criteria
* Baseline moderate and severe hepatic impairment (Child-Pugh Class B and C)
* Presence of uncontrolled hypertension, hypokalemia, or fluid retention
* History or presence of adrenocortical insufficiency
* Use of concomitant medications that are sensitive substrates for CYP2D6 with a narrow therapeutic index
* Use of strong CYP3A4 inducers

Subprotocol C only:

Inclusion criteria

* Subjects who are refractory to a novel antiandrogen therapy. Subjects must be ineligible for or refuse taxane therapy.
* Evidence of progressive disease, defined as 1 or more PCWG3 criteria: PSA level >/=1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart, nodal or visceral progression as defined by RECIST 1.1 with PCGW3 modifications, and/or appearance of 2 or more new lesions in bone scan Exclusion criteria
* History or evidence of interstitial lung disease or active, non-infectious pneumonitis
* Subjects on a prior PD-1 or PD-L1 inhibitor who experienced a grade 3 or higher immune-related adverse event prior to first day of dose

Subprotocol D only:

Inclusion criteria

* Subjects may have had novel hormonal therapies (NHT; eg, abiraterone, enzalutamide, apalutamide, or darolutamide) for prostate cancer, but no more than 1 NHT for metastatic prostate cancer
* Ineligible for or refuse taxane therapy

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Dose exploration only: Number of participants who experience dose limiting toxicities (DLTs) | Up to 3 years
  The analysis of all endpoints, unless noted otherwise, will be conducted on the Safety Analysis Set defined as all subjects that are enrolled and receive at least 1 dose of Acapatamab. The analysis of dose-limiting toxicity (DLT) will be conducted on the DLT Analysis Set defined as all subjects that are enrolled and receive at least 1 dose of Acapatamab with an evaluable DLT endpoint. If a single subject experiences more than 1 DLT it will be counted as 1.
  The DLT endpoint is evaluable if either:
  1) the subject experiences a DLT; or 2) the subject does not experience a DLT after receiving all planned doses within the 28-day DLT window in cycle 1.
Number of participants who experience one or more treatment-emergent adverse events (TEAEs) | Up to 3 years
Number of participants who experience one or more treatment-related adverse events | Up to 3 years
Number of participants who experience a clinically significant change in vital signs | Up to 3 years
Number of participants who experience a clinically significant change in clinical laboratory tests | Up to 3 years

SECONDARY OUTCOMES:
Objective response rate per response evaluation criteria in solid tumors (RECIST) 1.1 with prostate cancer working group 3 (PCWG3) modifications | Up to 3 years
Number of participants who experience circulating tumor cell (CTC) response | Up to 3 years
Number of participants who experience prostate-specific antigen (PSA) response rate | Up to 3 years
Duration of response | Up to 3 years
Overall survival (OS) | Up to 3 years
Progression-free survival | Up to 3 years
Time to progression | Up to 3 years
Time to subsequent therapy | Up to 3 years
Maximum plasma concentration (Cmax) | Up to 3 years
Minimum plasma concentration (Cmin) | Up to 3 years
Area under the concentration-time curve (AUC) | Up to 3 years
Accumulation ratio based on area under the concentration-time curve (AUC) | Up to 3 years
Half-life (t1/2) | Up to 3 years
Change from baseline in prostate-specific membrane antigen (PSMA)-positive tumor burden assessed using gallium (GA) 68-labelled PSMA-11 positron emission tomography/computed tomography (PET/CT) | Baseline up to 3 years
Change from baseline in prostate-specific membrane antigen (PSMA)-negative disease burden assessed using 18F-fluorodeoxyglucose (F-FDG) positron emission tomography/computed tomography (PET/CT) | Baseline to 3 years
Time to symptomatic skeletal events | Up to 3 years
Concentration of alkaline phosphatase | Up to 3 years
Concentration of lactate dehydrogenase (LDH) | Up to 3 years
Concentration of hemoglobin | Up to 3 years
Neutrophil-to-lymphocyte ratio | Up to 3 years
Concentration of N-telopeptide in the urine | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Irvine Medical Center, Orange, California
  - University of California San Francisco Mission Bay Campus, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- St Vincents Hospital Sydney, Darlinghurst, New South Wales, Australia
- Rigshospitalet, København Ø, Denmark
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain
- Sweden (3):
  - Skanes universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Akademiska sjukhuset, Uppsala
- Royal Marsden Hospital, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com